CLINICAL TRIAL: NCT03353090
Title: Incremental Diagnostic Utility of Systematic Double-bed SPECT/CT for Bone Scintigraphy in Initial Staging of Cancer Patients
Brief Title: Double-bed SPECT/CT for Bone Scintigraphy in Initial Staging of Cancer Patients
Acronym: DTOM
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: DTOM
Record Dates: First submitted 2017-11-10; First posted 2017-11-27 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Bone Metastases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bone scintigraphy is currently a reference test in the initial staging of cancer. Bone scintigraphy historically consists in a planar whole-body scintigraphy (WBS). SPECT/CT has been shown to dramatically reduce the proportion of inconclusive results and increase the specificity of bone scintigraphy. Therefore, in most of nuclear médicine centers, the usual protocol for staging of bone metastases consists in a whole-body planar acquisition followed, if needed, by a targeted SPECT/CT to characterize suspicious or equivocal uptakes seen on WBS. The aim of this study is to assess the incremental diagnostic utility of a systematic double-bed SPECT/CT acquisition for bone scintigraphy in initial staging of cancer patients compared with the conventional "WBS plus single-bed targeted SPECT/CT" strategy.

DETAILED DESCRIPTION:
Images are interpreted by two nuclear medicine physicians in a 3-step procedure and by consensus. Firstly,only WBS planar images are considered. Secondly, a single-bed SPECT/CT chosen based on planar images is used if WBS demonstrated any equivocal or suspicious uptake.

Finally, WBS and double-bed SPECT/CT images are used for interpretation.

A per-lesion, a per-anatomical region and a per-patient analysis is performed. At each step, lesions, regions and diagnostic conclusions are classified using a 3-level scale, as negative for malignancy, equivocal or suspicious for metastasis

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for bone scintigraphy for initial staging of biopsy proven malignancy.

Exclusion Criteria:

* monoclonal gammapathy
* patients under 18 years of age
* Technical issues not allowing a double-bed SPECT/CT acquisition
* double bed SPECT/CT acquisition not centered from the upper cervical spine to the proximal femora

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2016-12-10 (Actual); Study Completion 2016-12-10 (Actual)

PRIMARY OUTCOMES:
Diagnostic impact of a systematic double SPECT/CT as compared to a oriented single-bed SPECT/CT bone scintigraphy for staging of malignancies with bone scintigraphy | day 1

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France